CLINICAL TRIAL: NCT01347606
Title: Prospective Randomized Technical Study
Brief Title: Secured Thyroidectomy With Intraoperative Methylene Blue Using
Acronym: bluethyroid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SB Istanbul Education and Research Hospital (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: erhan aysan, Bezmialem Vakif University
Other Study IDs: 4-Aysan
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2010-01

CONDITIONS: Thyroid
Keywords: thyroid; secure; surgery; methylene; blue
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — thyroid tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
Thyroid surgery has potential risks. Intraoperative organ (such as parathyroides) extraction and vascular or neural (such as recurrent nervus) injuries are most important ones. This research is aim to prevention of these via intraoperative methylene blue using.

DETAILED DESCRIPTION:
Thyroid surgery has potential risks. Intraoperative organ (such as parathyroides) extraction and vascular or neural (such as recurrent nervus) injuries are most important ones. This research is aim to prevention of these via intraoperative methylene blue using. In the operation when thyroid lobes manipulated to medially, methylene blue will be sprayed to this area. Dying patternes of tissues (thyroid tissue, oparathyroid tissues, arteries, venules and neural structures) will ensure to identification the tissues.

ELIGIBILITY:
Inclusion Criteria:

* Thyroidectomy indicated patients

Exclusion Criteria:

* Recurrent disease
* Additional disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: thyroidectomy indicated patients
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: erhan aysan, Assoc. Prof., Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)